CLINICAL TRIAL: NCT06038058
Title: A Phase I Clinical Study of the Safety, Tolerability and Efficacy of BRY812 for Injection in Patients With Advanced Malignancies
Brief Title: A Study of BRY812 for Injection Alone in Subjects With Advanced Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BioRay Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRY812-ST-01
Record Dates: First submitted 2023-08-31; First posted 2023-09-14 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Advanced Malignancies
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BRY812 (Experimental)
  Interventions: Drug: BRY812 for injection

INTERVENTIONS:
Drug: BRY812 for injection — BRY812 for injection will be administered by intravenous drip, tentatively once per cycle spanning 3 weeks on D1 of each cycle until intolerable toxicity, disease progression, pregnancy, withdrawal of informed consent, death, study discontinuation or withdrawal from the study. The dose of each administration will be calculated based on the weight measured prior to such administration. The dosing regimen (dosing frequency and interval) for subsequent study may be adjusted based on prior data. The intravenous drip should last for ≥ 90 min for the first dose and may be adjusted to ≥ 30 min for subsequent doses if the first dose is tolerable.

SUMMARY:
This is a Phase I, multicenter, open-label, single-arm and first-in-human clinical study of BRY812 for injection. The study objectives are to evaluate the safety, tolerability, pharmacokinetic profile, anti-tumor activity and immunogenicity of BRY812 for injection in patients with advanced malignancies.

Patients will receive treatment every 3 weeks until intolerable toxicity, disease progression, pregnancy, withdrawal of informed consent, death, study discontinuation, or withdrawal from the study.

ELIGIBILITY:
Inclusion Criteria:

* (1) Subjects who voluntarily sign the informed consent form, understand the nature, objectives, and procedure of the study and are able to complete the study according to the protocol;
* (2) Male or female patients, ≥ 18 years of age (based on the date of signing the informed consent form);
* (3) In Phase Ia: patients must have advanced solid tumors confirmed by histopathology and/or cytology, who have failed to respond to standard-of-care (disease progression after treatment) or who could not tolerate standard-of-care, or who could not obtain effective standard-of-care or for whom there was no effective standard-of-care available; (Note: the patient population and inclusion criteria in phase Ib will be determined according to the data of phase Ia);
* (4) According to RECIST v1.1 (Response Evaluation Criteria in Solid Tumors), there is at least 1 measurable lesion;
* (5) Eastern Cooperative Oncology Group (ECOG) Status 0 to 1;
* (6) Adequate organ and bone marrow function (no treatment with cells, growth factors, or transfusions within 14 days prior to the first administration), as defined below:

  1. Hematology: absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count (PLT) ≥ 100 × 109/L, hemoglobin (HGB) ≥ 90 g/L;
  2. Liver function: serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN) (except for subjects with Gilbert syndrome, TBIL ≤ 2 × ULN in patients with liver cancer or liver metastases), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (in patients with liver cancer or liver metastases, ALT or AST ≤ 5 × ULN);
  3. Renal function: creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance (CrCL) (based on Cockcroft-Gault equation) ≥ 60 mL/min;
* (7) Expected survival ≥ 12 weeks;
* (8) Female subjects with fertility potential must test negative for serum human chorionic gonadotropin (HCG) before they are enrolled in the study. Female subjects with fertility potential or male subjects who have a female partner must agree to maintain no pregnancy plan and take effective contraceptive measures such as condoms from the signing of ICF to 6 months after the last dose of study drug (see Annex 1 for details); females are considered fertile from menarche to menopause (at least 12 months without menstruation) unless they are permanently infertile (through hysterectomy, bilateral salpingectomy, or bilateral oophorectomy).

Exclusion Criteria:

* (1) Subjects who have previous severe hypersensitivity to BRY812 or known hypersensitivity to any component or excipient of the study drug;
* (2) Subjects who have previously received drugs which target LIV-1;
* (3) Subjects who have any active infection requiring systemic therapy by intravenous infusion within 2 weeks prior to the first dose of study drug;
* (4) Subjects who have previous or current presence of two or more primary tumors (excluding cured cervical carcinoma in situ, basal cell carcinoma, or squamous cell carcinoma of the skin, and other tumors that have been stable for more than 5 years after treatment);
* (5) Subjects who have symptoms of active central nervous system metastases, except those with brain parenchymal metastases assessed as stable by the investigator based on the following conditions:

  1. No seizures within > 12 consecutive weeks with or without the treatment of antiepileptic drugs;
  2. Glucocorticoids are not required;
  3. Two consecutive MRI scans (at least 4 weeks apart) show a stable state on imaging;
  4. Asymptomatic inactive brain metastases are newly identified where two consecutive MRI scans (at least 4 weeks apart) show a stable state on imaging;
  5. The conditions remain stable and asymptomatic for more than 1 month after treatment;
* (6) Subjects with serious cardiovascular and cerebrovascular diseases and lung diseases, including but not limited to:

  1. Stroke, intracranial hemorrhage, unstable angina pectoris, congestive heart failure (NYHA class III-IV), myocardial infarction, severe arrhythmias (such as sustained ventricular tachycardia and ventricular fibrillation), congenital long QT syndrome, torsade de pointes, and symptomatic pulmonary embolism within 6 months before enrollment;
  2. Uncontrolled hypertension (at least 2 consecutive measurements of systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg);
  3. Echocardiogram (ECHO) or multigated acquisition scan (MUGA) shows left ventricular ejection fraction (LVEF) < 50%;
  4. During the screening period, the mean corrected (by Fridercia's formula) QT interval on three consecutive electrocardiograms is prolonged (> 450 ms in males and > 470 ms in females);
  5. Subjects who have interstitial lung diseases, severe impaired lung function, severe pulmonary fibrosis, radiation pneumonitis, and other lung diseases assessed by the investigator as clinically significant;
* (7) Subjects who have active gastrointestinal bleeding or severe intestinal obstruction;
* (8) Subjects who have undergone major surgery within 4 weeks prior to the first dose of study drug or are expected to be performed during the study;
* (9) Subjects who have a history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* (10) Subjects who have bleeding tendency or are receiving thrombolytic or anticoagulant therapy;
* (11) Subjects who have used strong inhibitors or substrates of CYP3A4 and/or Pgp within 4 weeks before the first dosing or within 5 half-lives of the used drug (whichever is shorter), or who have received anti-tumor therapy or participated in other clinical studies and used other study drugs, including chemotherapy, targeted therapy, immunotherapy, biotherapy (tumor vaccines, cytokines, or growth factors for cancer control), etc.; or who have received prepared slices of Chinese crude drugs or Chinese patent medicines as anti-tumor treatment within 1 week before the first dose of study drug;
* (12) Subjects who have received radiation therapy, including abdominal palliative stereotactic radiotherapy, within 4 weeks prior to the first dose of study drug (non-abdominal palliative stereotactic radiotherapy within 2 weeks prior to the first dose);
* (13) Toxicity of previous antineoplastic therapy does not resolve to grade ≤ 1 as defined by NCI-CTCAE v5.0 (except for asymptomatic abnormal laboratory findings considered by the investigator, such as elevated ALP, hyperuricemia, elevated blood glucose, etc.; except for toxicity with no safety risk determined by the investigator , such as alopecia, pigmentation, etc.);
* (14) Subjects who have been vaccinated with a live vaccine within 4 weeks before the first dose, or who intend to be vaccinated with a live vaccine during the study;
* (15) Subjects who have received more than 1 week of treatment with systemic corticosteroids (methylprednisolone > 10 mg/day or an equivalent dose of other similar drug) within 2 weeks prior to the first dose of study drug;
* (16) Subjects who have used immunosuppressants within 2 weeks prior to the first dose or once had active autoimmune diseases or had a prior history of autoimmune diseases;
* (17) Subjects who test positive for Hepatitis B surface antigen (HBsAg) with HBV DNA beyond the normal range; or subjects who test positive for hepatitis B core antibody with HBV DNA beyond the upper limit of normal, but do not agree to regular DNA testing during treatment and follow-up, or do not agree to receive antiviral therapy; subjects who test positive for hepatitis C virus (HCV) antibody and HCV RNA; subjects who are seropositive for human immunodeficiency virus (HIV); subjects who have syphilis and need to receive systemic treatment;
* (18) Subjects who have any mental or cognitive disorders that may limit their understanding and execution of the informed consent form;
* (19) Subjects who are pregnant or breastfeeding;
* (20) Subjects who plan to donate sperm after signing the informed consent form and throughout the study period, or within 6 months after the last dose of the study drug;
* (21) Subjects who are not eligible for enrollment or may not be able to complete the study due to other reasons by the investigator's assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From Day 1 to 30 days after last dose; approximately 2 years
  An AE is any untoward medical occurrence in a patient or clinical investigational subjct administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Incidence of laboratory abnormalities | From Day 1 to 30 days after last dose; approximately 2 year
  To be summarized using descriptive statistics
Maximum Tolerated Dose (MTD) of BRY812 for injection | From the first dose to the last dose；approximately 2 year
  Maximum Tolerated Dose (MTD) of BRY812 for injection
Recommended phase II dose (RP2D) of BRY812 for injection | From the first dose to the last dose；approximately 2 year
  Recommended phase II dose (RP2D) of BRY812 for injection
Incidence of dose-limiting toxicity (DLT) | Through 21 days after first dose
  Incidence of dose-limiting toxicity (DLT)

SECONDARY OUTCOMES:
Objective response rate (ORR) | Through 1 month following last dose; approximately 2 years
  ORR is defined as the proportion of patients with complete response (CR) or partial response (PR) per RECIST v1.1.
Progression-free survival (PFS) | Up to approximately 3 years
  PFS is defined as the time from start of study treatment to first documentation of tumor progression (clinical progression or PD per RECIST v1.1).
Overall survival (OS) | Up to approximately 3 years
  OS is defined as the time from start of study treatment to date of death due to any cause
Duration of response (DOR) | Up to approximately 3 years
  DOR is defined as the time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of tumor progression (clinical progression or progressive disease (PD) per RECIST v1.1)
Pharmacokinetic assessment | Through 18 weeks after dosing
  The concentrations of BRY812, total antibody and free monomethyl auristatin E (MMAE) in blood will be determined.
Immunogenicity assessment | Through 18 weeks after dosing
  The anti-drug antibody (ADA) of BRY812 in the blood is detected, and the antibody titer of ADA-positive patients is further detected according to the situation, and whether they have neutralizing antibody (NAb) is detected if necessary.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital，Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No